CLINICAL TRIAL: NCT00467753
Title: Oxcarbazepine Versus Placebo in Childhood Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Sherie Novotny, M.D., Assistant Professor, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0220055339
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Autism
Keywords: Irritability; Functional Ability; Aggression; Mood Instability
MeSH Terms: conditions — Autistic Disorder; Aggression | interventions — Oxcarbazepine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxcarbazepine (Experimental): Oxcarbazepine is the active drug to be given to subjects in the experimental arm
  Interventions: Drug: Oxcarbazepine
- Sugar Pill (Placebo Comparator): Patients are given either active or inactive intervention.
  Interventions: Other: Placebo/sugar pill

INTERVENTIONS:
Drug: Oxcarbazepine — Oxcarbazepine is available in a 300mg/5ml solution. Dosage will start at 150 mg (2.5ml) at night for 3 days and will be increased to 150 mg in the am and pm. For children who are able to tolerate the 150 mg BID dose, the oxcarbazepine will be increased to 300 mg at night and 150 mg in the morning for 3 days and 300 mg BID for the next week. The children will remain on this dose until week 3, at which time if they are tolerating the medication and do not have a Clinical Global Improvement Scale (CGI) of 1 (very much improved) they will be increased to 600 mg twice a day in a method similar to the above increases. After week 4, the child will remain on the same stable dose.
  Other Names: Trileptal
  Arms: Oxcarbazepine
Other: Placebo/sugar pill — Dosage similar to active drug
  Arms: Sugar Pill

SUMMARY:
The proposed study is designed to assess the effectiveness of treatment with Oxcarbazepine vs. placebo in childhood/adolescent autism. This is a twelve-week study involving twenty subjects between the ages of five and seventeen with a diagnosis of autism.

DETAILED DESCRIPTION:
The proposed study is designed to assess the effectiveness of treatment with Oxcarbazepine vs. placebo in childhood/adolescent autism. This is a twelve-week study involving twenty subjects between the ages of five and seventeen with a diagnosis of autism. Subjects will receive a psychiatric and medical evaluation by the study psychiatrist to see if she/he has any psychiatric or medical illnesses that would interfere with their ability to participate in this study. These evaluations may take up to an hour to complete. In addition, subjects will be asked to participate in a psychiatric interview designed to determine the child's diagnosis and current problem areas. The subject's parent will also be asked to fill out psychiatric questionnaires. The interview and questionnaires may take up to 4 hours to complete.

ELIGIBILITY:
Inclusion Criteria:

* Subject has autism.
* Subject is between five and seventeen years of age
* Subject is not hospitalized.

Exclusion Criteria:

* Subject has been diagnosed with a psychopathic disorder or a mood disorder, including depression or bipolar disorder.
* Subject has displayed self-injurious behavior.
* Subject has an active seizure disorder or epilepsy.
* Subject has an unstable medical illness.
* Subject has undergone brain injury.
* Subject has a history of diabetes.
* Subject has a history of prior treatment with oxcarbazepine of 600 mg/day for 6 weeks.
* Subject has used other study drugs within the previous 30 days.
* Subject is a pregnant female or unwilling to use acceptable contraception if sexually active.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2006-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherie L. Novotny, M.D, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- Child and Adolescent Psychiatry at the University Behavioral Healthcare Building, UMDNJ-RWJMS, Piscataway, New Jersey, United States

REFERENCES:
- See also: University Behavioral Healthcare official site — http://ubhc.umdnj.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study was ineffective resulting in only 5 patients recruited, and 0 completers.
Groups:
- Oxcarbazepine: Oxcarbazepine is the active drug to be given to subjects in the experimental arm
  Oxcarbazepine : Oxcarbazepine is available in a 300mg/5ml solution. Dosage will start at 150 mg (2.5ml) at night for 3 days and will be increased to 150 mg in the am and pm. For children who are able to tolerate the 150 mg BID dose, the oxcarbazepine will be increased to 300 mg at night and 150 mg in the AM for 3 days and 300 mg BID for the next week. The children will remain on this dose until week 3, at which time if they are tolerating the medication and do not have a CGI of 1 (very much improved) they will be increased to 600 mg twice a day in a method similar to the above increases. After week 4, the child will remain on the same stable dose.
- Sugar Pill: Placebo : Dosage similar to active drug
Period: Overall Study
Arm/Group | Oxcarbazepine | Sugar Pill
Started | 3 | 2
Completed | 0 | 0
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: 5 patients started in the study, 2 dropped out after 1-2 weeks , 3 were lost to follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxcarbazepine | Sugar Pill | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (2) | 12.5 (3) | 9.8 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Vineland Adaptive Behavior Scales
Description: The Vineland Scale is a semi-structured informant interview that assesses subjects' functioning. It is administered to a caretaker/family member. The scale has been revised and standardized in all populations. This scale has been found to assess social deficits in autism and strengths in daily living skills. Items are classified under four major adaptive domains: communication, daily living skills, socialization and motor skills. The items are scored 0-2 (yes/sometimes/never). Each domain is summed, and the domain scores are converted to standardized scores. The normative score is 100, with standard deviation of 15. The standardized score is used in this study. A higher score (above 100) means better adaptive behavior. Minimum value is 0, maximum value is infinity.
Time Frame: Evaluated during Baseline and Termination
Population: Zero participants analyzed
Arm/Group | Oxcarbazepine | Sugar Pill
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Aberrant Behavior Checklist
Description: Aberrant Behavior Checklist (ABC)-Community Version (Irritability Subscale) (Aman et al. 1985). It is designed to objectively identify five behavior subscales through observation by the primary caregiver. The five behavior subscales include (ranges show no problem to severe problem): irritability (range 0-45), lethargy (range 0-48), stereotypy (range 0-21), hyperactivity range 0-48), and inappropriate speech (range 0-12), all possible signs and symptoms of affective instability in autistic individuals (Lainhart & Folstein, 1994). Improvement is shown with scores decreasing over time. Total score is not used. Inter-rater reliability for the ABC-CV is moderate to high across subscales with a mean of .63. Test-retest reliability correlations are .98 -Irritability, .99 -Lethargy, .98 -Stereotypy, .98 -Hyperactivity, and .96 -Inappropriate Speech. The ABC will be filled out by an informant (teacher/parent), and then reviewed by the IE. Administration time is approximately 10 minutes.
Time Frame: Bi weekly
Population: There were not enough participants in this study to analyze results.
Arm/Group | Oxcarbazepine | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Autism Diagnostic Observation Schedule
Description: The Autism Diagnostic Observation Schedule is primarily used as a diagnostic tool providing a standardized assessment for observation of social and communicative behavior in children and adults. It is composed of four modules for assessing children/adults of varying language ability (Module 1 for nonverbal individuals, to Module 4 fluent individuals). The instrument provides a series of structured and semi-structured presses for social interaction and communication, which are then scored. The scores are 0 (no behavior) to 3 (markedly abnormal). Subcategories are Language/communication, 8 scores, Social interaction, 12 scores, Stereotyped Behavior/restricted interests, 4 scores and Play, 2 scores, as well as other behavior, 3 scores. The maximum score is 87, minimum is 0, with cutoff scores to determine diagnosis. Higher scores indicate a more severe behavioral disorder.
Time Frame: Evaluated during Baseline and Termination
Population: There were not enough participants to analyze the data in this study.
Arm/Group | Oxcarbazepine | Sugar Pill
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Clinical Global Impression Improvement (CGI-AD)
Description: Clinical Global Impression Improvement (CGI)-AD (Guy, 1976). This is a standard rating scale with 7-point global severity and change scales which has been modified for Autistic Disorder. A rating of 2 is given when there is a substantial reduction in symptoms so that a treating clinician would be unlikely to change treatment. A rating of 1 is reserved for patients who become virtually symptom-free. A rating of 3 (minimally improved) on the CGI is defined as slight symptomatic improvement that is not deemed clinically significant. Administration time is approximately 2 minutes.
Time Frame: Administered weekly Administered weekly
Population: There were not enough participants in this study to analyze results.
Groups:
- Oxcarbazepine; Placebo/Sugarpill: There were not enough participants in this study to analyze results.
Arm/Group | Oxcarbazepine | Placebo/Sugarpill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: OVER THE ONE YEAR OF THE STUDY
Description: Irritability due to weaning from effective medication.
Arm/Group | Oxcarbazepine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxcarbazepine (N=3) | Sugar Pill (N=2)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) — Two children became irritable due to being off of their previous medications and could not continue in the study. One was on active and dropped in week 4 the other dropped at week 1.

LIMITATIONS AND CAVEATS:
Patients became more irritable coming off of previous medication and were unable to tolerate monotherapy with the medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No